CLINICAL TRIAL: NCT07026539
Title: Effect of Treatment With Finerenone on Cardio-Renal Target Organ Damage in Patients With Type 2 Diabetes - A Randomized Trial
Brief Title: Effect of Treatment With Finerenone on Cardio-Renal Target Organ Damage in Patients With Type 2 Diabetes.
Acronym: FineCaRe
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20235044465800; 2023-504446-58-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Chronic Kidney Disease Due to Type 2 Diabetes Mellitus; Cardiovascular Diseases
Keywords: Mineralocorticoid receptor antagonist (MRA); Type 2 diabetes; Chronic kidney disease; Diabetic complications; finerenone
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Renal Insufficiency, Chronic; Diabetes Complications | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Finerenone (active) (Experimental)
  Interventions: Drug: Finerenone (BAY 94-8862)

INTERVENTIONS:
Drug: Finerenone (BAY 94-8862) — Patients with an eGFR of 25-60 ml/min/1.73m2 will receive an initial dose of 10 mg finerenone/placebo once daily and those with an eGFR of at least 60 ml/ in/1.73m2 will receive an initial dose of 20 mg finerenone/placebo once daily. From 4 weeks the target dose is 20 mg finerenone/placebo once daily. An increase in dose from 10 to 20 mg once daily will be encouraged after 4 weeks provided the plasma potassium level is 4.8 mmol/L or less and the eGFR stable. If eGFR is reduced with >30 % compared to the previous measurement, we will not increase the dose of finerenone/placebo. Plasma potassium and eGFR will be measured 4 weeks after any initiation, re-start or increase in dose. A decrease in dose from 20 to 10 mg is allowed at any time after initiation of finerenone or placebo. Patients in the placebo group will undergo sham adjustment of the dose. Finerenone or placebo will be withheld if potassium concentrations exceed 5.5 mmol/L and restarted if potassium levels fall to 5.0 mmol/L
  Arms: Finerenone (active)
Drug: Placebo — Placebo tablets matching BAY94-8862 are administered orally.
  Arms: Placebo

SUMMARY:
The global prevalence of diabetes is increasing substantially. Around 40 % of patients with type 2 diabetes develop chronic kidney disease. Diabetic kidney disease is the leading cause of kidney failure, it is closely linked to cardiovascular disease and heart failure and is associated with a threefold increase in all-cause mortality and a 16-year loss in life expectancy.

In large clinical trials, the novel drug finerenone has shown to lower the risk of chronic kidney disease progression and improve the cardiovascular outcome for patients with type 2 diabetes and chronic kidney disease. However these trials did not not reflect current standard-of-care for patients with type 2 diabetes and chronic kidney disease, as only a minority (6.7 %) received an SGLT2-I - a treatment that has been considered standard-of-care for these patients since 2022.

The FineCaRe study aims to investigate the effect of treatment with finerenone in combination with an SGLT2-I on albuminuria and left ventricular mass in patients with type 2 diabetes and chronic kidney disease.

The investigators will perform a 26-week investigator-initiated, single-center, placebo-controlled, double-blinded randomized clinical trial. After screening and inclusion, participants will be randomized 1:1 to either finerenone or placebo treatment. Outcomes will be assessed at baseline, during and after 26 weeks of treatment.

The primary goal of the FineCaRe study is to acquire new knowledge that may help in preventing kidney failure in diabetic patients. With this project the investigators aim to contribute to the understanding of which disease mechanisms in the kidneys and heart that can be targeted in diabetic patients with kidney disease. This could hopefully provide better opportunities for preventing chronic kidney disease and kidney failure.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Diagnosis of type 2 diabetes according to the World Health Organization definition.
* Current treatment with a SGLT2-I1 at maximally tolerated dose.
* Current treatment with an ACE inhibitor or an ARB1 at maximally tolerated dose.
* Plasma potassium level of 4.8 mmol/L or less at the time of screening.
* CKD defined as eGFR ≥25 ml/min/1.73 m2 and albuminuria (UACR between 30-5000 mg/g).
* Speak and understand Danish fluently.

Exclusion Criteria:

* Inability to give informed consent.
* Severe renal disease with eGFR <25 ml/min/1.73m2.
* Severe hepatic disease (plasma ALAT above 3 x upper limit of normal).
* Active cancer diagnosis other than basal cell carcinoma.
* Treatment with systemic steroids at time of randomization.
* Bariatric surgery within 2 years or other gastrointestinal surgeries that induce chronic malabsorption.
* Alcohol or drug abuse within 3 months of informed consent that would interfere with trial participation or any ongoing condition leading to decreased compliance with study procedures or study drug intake.
* Chronic or acute pancreatitis.
* Pregnancy or breastfeeding (see pregnancy below).
* Poorly controlled medical condition, e.g. congestive heart failure (New York Heart Association III-IV or EF ≤ 40%), recent (within 3 months) stroke or acute myocardial infarction or any other condition that in the opinion of the investigator will put the trial participant at risk if participating in the trial.
* Allergy to finerenone or any of the excipients contained in the drug.
* Current systemic treatment with strong inhibitors of CYP3A4 (e.g. itraconazol, ketoconazole, ritonavir, cobicistat, clarithromycin) or strong inducers of CYP3A4 (e.g. rifampicin, carbamazepine, phenytoin, phenobarbital).
* Current treatment with other MRAs (e.g. spironolactone, eplerenone etc.).
* Patients with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose- galactose malabsorption.
* Addison's disease.
* Contraindications to MRI.
* Previous renal or heart transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular mass measured by non-contrast cardiac MRI of the heart | From the baseline visit at week 0 to the end of treatment at week 26.
Change in albuminuria measured by a urinary albumin-to-creatinine ratio (UACR) in morning spot urine samples (first morning voids). | From the baseline visit at week 0 to the end of treatment at week 26.

SECONDARY OUTCOMES:
Change in the rate of myocardial fibrosis (extracellular cardiac volume - ECV %) measured by MRI of the heart using gadolinium-containing contrast. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in the rate of myocardial fibrosis measured by non-contrast T1-mapping using MRI of the heart. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in left ventricular ejection fraction (EF), left ventricular and atrial volumes measured by non-contrast MRI of the heart. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in thoracic aortic wall volume (TWV) measured by MRI of the heart. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in the rate of pulse wave velocity in the aorta measured by non-contrast MRI of the heart. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in arterial stiffness assessed as cf-PWV. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in 24-hour blood pressure. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in inflammatory and fibrotic biomarkers related to CVD measured in blood and urine. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in measured glomerular filtration rate (mGFR) assessed by injection of a tracer. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in eGFR slope including all available outpatient eGFR measured a) from before treatment to last day of treatment b) from 4 weeks after treatment initiation to last day after treatment. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in UACR by repeated measures analysis including all available outpatient UACR measurements from before treatment to the last day after treatment. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in markers of the RAAS measured in blood and urine. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in inflammatory and fibrotic biomarkers related to CKD (e.g. markers of renal tubule damage) measured in blood and urine. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in kidney microstructure and fibrosis assessed as changes in T1-mapping and changes in the rate of ADC-values of diffusion-weighted MRI of the kidneys using non-contrast MRI. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in renal oxygenation assessed by BOLD MRI and change in renal perfusion with a pseudo continuous arterial spin labeling (pCASL), both non-contrast MR techniques | From the baseline visit at week 0 to the end of treatment at week 26.
Change in kidney size measured by a Dixon water/fat sequence MRI, a non-contrast MRI technique. | From the baseline visit at week 0 to the end of treatment at week 26.

OTHER OUTCOMES:
Change in retinal thickness assessed with Optical Coherence Tomography (OCT). | From the baseline visit at week 0 to the end of treatment at week 26.
Change in retinal oxygenation measured by oximetry. | From the baseline visit at week 0 to the end of treatment at week 26.
Change in the transcriptomic, proteomic, and/or metabolomic profile in plasma and urine. Furthermore, to test if possible changes can be related to pathways involved in and/or serve as biomarkers of the progression of cardiovascular and/or kidney disease | From the baseline visit at week 0 to the end of treatment at week 26.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during the described study will not be publicly available due to privacy and ethical restrictions. Interested parties can request access to deidentified data or anonymised study reports by submitting a request to the primary investigator, provided that the necessary data protection agency and ethical committee approvals are given, in compliance with relevant legislation.